CLINICAL TRIAL: NCT07155811
Title: Prospective, Single-center, Clinico-biological Cohort Evaluating the Automated VIDAS STIMM T Test in Patients With Advanced/Metastatic Solid Tumors Treated With Standard Immunotherapy
Brief Title: Lymphocyte Function Testing in Immuno-oncology
Acronym: T-ECHNICO
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Leon Berard (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: ET24-155 T-ECHNICO; EU number (Other: 2024-A01300-47)
Record Dates: First submitted 2025-08-20; First posted 2025-09-04 (Actual); Last update posted 2025-09-04 (Actual); Status verified 2025-08

CONDITIONS: Immunotherapy; Advanced Solid Tumor Malignancies

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cohorte A: Immunothérapie sans chimiothérapie concomitante (Active Comparator): Immunotherapy without concurrent chemotherapy
  Interventions: Diagnostic Test: test immunitaire fonctionnel automatisé VIDAS® STIMM™ T RUO
- Cohorte B : Immunothérapie avec chimiothérapie concomitante (Active Comparator): Immunotherapy with concurrent chemotherapy
  Interventions: Diagnostic Test: test immunitaire fonctionnel automatisé VIDAS® STIMM™ T RUO

INTERVENTIONS:
Diagnostic Test: test immunitaire fonctionnel automatisé VIDAS® STIMM™ T RUO — The functional assessment of T lymphocytes is based on the use of the VIDAS® STIMM™ T RUO test, which will be performed on freshly collected whole blood in lithium heparin tubes without gel separators. Blood samples will be sent to the Immunology Laboratory at E. Herriot Hospital (Prof. Guillaume Monneret). T lymphocytes will be stimulated ex vivo for 3.5 hours (non-antigen-dependent stimulation by PHA) on the VIDAS®3 automated system (bioMérieux).
  The automated system then performs a assay (immunofluorescence technique) to quantify the concentrations of IFN-γ in the supernatant of each sample. The entire process is automated, and results are obtained within 4 hours.

SUMMARY:
Several studies have shown that the presence and levels of IFN-γ may correlate with better responses to immunotherapy. Higher baseline levels of IFN-γ and an increase in its production during treatment have been associated with better clinical outcomes in patients receiving immunotherapy such as anti-PD-1/PD-L1 or anti-CTLA4.

To date, there is no simple, rapid, automated, and standardized test to assess T-cell functionality and quantify the level of immunosuppression in individual patients. To address this medical need, bioMérieux has developed the VIDAS® STIMM™ T RUO automated functional immune test, which can determine a patient's immune status by measuring IFN-γ production by T lymphocytes after stimulation by a mitogen in approximately four hours without human intervention. The aim of this study is to evaluate whether the amount of IFN-γ produced by T lymphocytes, as measured by an automated VIDAS® STIMM™ T functional immune test, correlates with disease progression in patients with advanced/metastatic solid tumors treated with standard immunotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Male or female aged 18 years or older with a confirmed diagnosis of solid tumors (any type of tumor) in advanced or metastatic stages
* Patients who are due to start standard treatment with anti-PD1, anti-PDL1, or anti-CTLA4 (combinations of ICIs are permitted) at the Léon Bérard Center:

  * Cohort A: ICI without concomitant chemotherapy
  * Cohort B: ICI with concomitant chemotherapy
* Patients who have understood, dated, and signed the consent form for this study before undergoing any protocol-specific procedures.
* Patients affiliated with or covered by a social security system.

Exclusion Criteria:

* Patients to be treated with immunotherapy in combination with targeted therapy.
* Patients treated with chemotherapy within the last 21 days prior to D1 of immunotherapy
* Pregnant or breastfeeding patients.
* Patients with other known cancers that are progressing or requiring the initiation of another treatment.
* Patients with psychological, family, geographical, or social circumstances that, in the investigator's judgment, could potentially prevent the signing of an informed consent form and/or compliance with study procedures.
* Patients in one or more of the following situations: subject to legal protection measures, deprived of liberty by judicial or administrative decision, receiving psychiatric care, admitted to a health or social care facility for purposes other than research

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-09-23 (Estimated); Primary Completion 2025-09-23 (Estimated); Study Completion 2025-09-23 (Estimated)

PRIMARY OUTCOMES:
Main objective of the study | up to 12 months
  Evaluate whether there is a correlation between T-cell function and radiological response under standard immunotherapy

IPD SHARING:
Plan to Share IPD: No